CLINICAL TRIAL: NCT04154839
Title: Pilot Study: Epidemiological Survey and Genetic Analysis of Patients With Atopic Dermatitis in Hong Kong
Brief Title: Epidemiological Survey and Genetic Analysis of AD Patients in Hong Kong
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr. Mandy Chan, Clinical Assistant Professor, The University of Hong Kong
Other Study IDs: UW 19-417
Record Dates: First submitted 2019-10-29; First posted 2019-11-07 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Atopic Dermatitis; Genetic Skin Disease; Eczema
Keywords: Atopic dermatitis; Genetics; Eczema; Epidemiology
MeSH Terms: conditions — Dermatitis, Atopic; Skin Diseases, Genetic; Eczema

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample in K2EDTA and SST tubes and/or buccal swab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Atopic dermatitis group: Number of subjects in atopic dermatitis group 0 - < 6 years : 50 subjects 6 - <12 years : 50 subjects 12 - <18 years : 50 subjects Adult (>= 18 years) : 150 subjects Total no. of cases: 300 cases
- Control group: >= 40 yrs : 150 subjects

SUMMARY:
This is a joint research study between The Hong Kong Polytechnic University (PolyU) and The University of Hong Kong (HKU) as titled above. In view of the increasing prevalence of atopic dermatitis (AD), the lack of complete epidemiology data on childhood and adult AD in Hong Kong and the lack of complete understanding on the genetic and environmental factors associated with it, the purpose of this study to carry out an epidemiology and genetic study that targets AD patients within the local Hong Kong population.

The investigators will search for new AD-associated genetic variants that are related to the local population and believe that the genetic profiles that arise from this project will form an important basis for the future management and treatment of AD, such as disease-risk screening strategy and therapeutic target development.

DETAILED DESCRIPTION:
Atopic dermatitis (AD), atopic eczema or eczema, is a very common, highly pruritic chronic inflammatory skin disorder. The intense itching, sleep disturbance, coupled with visible rashes, causes immense physical, psychological, economical and social implications. Not only does it impact on the quality of life of the patient, caregivers are also often affected. AD can manifest during childhood, adolescence or adulthood. Those with childhood-onset AD can go into remission during puberty and adolescence, or persist into adulthood. The natural course of AD is generally intermittent and seasonal, with phases of latency and exacerbation. AD is a heterogeneous condition with typical manifestations of other allergic disorders, but clinically, AD is defined as a single disorder. It is impossible to propose a definitive gold standard for the diagnosis of AD due to its heterogeneity. The most widely used diagnostic criteria is the Hanifin and Rajka criteria with reported sensitivity and specificity of 87.9-96.0% and 77.6-93.8% respectively.

SCORAD (SCORing Atopic Dermatitis) is one of the common clinical tools for assessing the extent and severity of AD. However, the molecular pathogenesis behind AD is still not fully understood, and the condition is not yet curable. The prevalence of AD is on the rise worldwide especially among industrialized countries, with an overall prevalence of around 15-30% among children and 0.3-14% among adults. In China, the overall prevalence of childhood/adolescent onset AD and adult onset AD are estimated at around 3.1% and 4.6% respectively. Variability in the overall prevalence is most likely due to non-standardized diagnostic criteria applied across various studies, originally designed only for childhood-onset AD. In Hong Kong, the epidemiological data on AD is incomplete and only childhood-onset AD was studied. Given that a significant proportion of AD patients belong to the adult-onset group, it is important to determine accurately the epidemiology of both childhood-onset and adult-onset AD groups in Hong Kong.

Recent evidence has also suggested that AD as a whole is attributed to a mixture of environmental and genetic factors, as AD has been shown to cluster in families and demonstrate high concordance in monozygotic twins. Various research studies have been conducted to identify environmental risk factors worldwide. In Hong Kong, Hon et al. from the Department of Pediatrics at The Chinese University, conducted a cohort study following up 82 children with AD for 10 years, and found that risk factors are often related to urbanization and exposure to aeroallergens. However, it is unclear whether both genetic predisposition and environmental factors also play a role in adult-onset AD group.

Apart from environmental factors, researchers have used different methods, such as genome-wide association study (GWAS), to search for genetic variations associated with childhood-onset AD. Several large-scale GWAS and candidate gene studies have been conducted on children-onset AD around the world to search for genetic risk factors using single nucleotide polymorphisms (SNPs). In China, Sun et al. performed the first GWAS in China in 2011 among 1012 children cases and 1362 adult controls of Southern Chinese to search for common genetic variants using Illumina Human 610-Quad Beadchips, followed by three replication studies among Northern Chinese, Southern Chinese and German cases and controls using MassArray and TaqMan assay. Although no robustly replicated SNPs have been identified across all GWAS and candidate gene studies, the commonest associated genetic variants, are related to the different loss-of-function mutations that encodes for the filaggrin (FLG). Filaggrin is a filament-aggregating protein that binds keratin fibers in epithelial cells. The loss-of-function mutations in FLG leads to enhanced transepidermal water loss, ichthyosis, penetration of foreign antigens, and subsequent sensitization . Other genetic variants, related to defective immune pathway and impaired skin barrier function have also been suggested in the past as risk factors for pathogenesis of AD. Despite this, there is currently no published data comparing genetic variants between adult-onset and children-onset AD groups. In addition, GWAS study in AD patients has not been conducted in Hong Kong.

The study will be conducted in compliance with local Institutional Review Board (IRB) and Good Clinical Practice (GCP).

ELIGIBILITY:
Inclusion Criteria:

Normal controls (Recruited in Poly U)

* Aged more or equal to 40 [Age of 40 is chosen as an arbitrary cutoff because studies had shown that the peak incidence among adult-onset AD cases occurs at age 20-40 years (Silvestre Salvador et al., 2017). Controls have been chosen more or equal to 40 years of age as they would likely have developed AD by the age of 40.
* Subjects that do not have a history of AD, personal history and family history of AD including first-, second-, and third-degree relatives;
* Subjects without a personal history and/or family history of other allergic and atopic disorders such as autoimmune diseases, skin disorders and systemic diseases.
* Born in Hong Kong and Chinese-Han

AD cases (Recruited from QMH and TWH)

* Patients have to be clinically diagnosed by a qualified dermatologist on the basis of a skin examination diagnosed according to Hanifin and Rajka criteria.
* Children cases should be aged < 18 at the time of recruitment and adult cases should be aged 18 at the time of recruitment;
* Born in Hong Kong and Chinese-Han

Exclusion Criteria:

* Non-Chinese or non-local case and control subjects;
* Either of the parents are non-Chinese;
* Case and control subjects who do not speak or understand Cantonese or Chinese;
* Age <40 for control subjects;
* Subjects who are pregnant;
* Unable to provide signed informed consent.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: For AD cases:
  Chinese-Han AD subjects who was born in Hong Kong
  For Control:
  Chinese-Han subjects who was born in Hong Kong aged more or equal to 40 Years
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2019-07-12 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Significant SNPs | through study completion, an average of 1 year
  The significant single nucleotide polymorphisms (SNPs) between control group and different AD case subgroups (different age of onset, different AD severity, different relapsing status), Cochran-Armitage trend test will be used to assess statistical significance of the association with each SNP, and Mantel-Haenszel method for two 2 × 2 allele frequency tables will be used to assess association of SNPs on chromosome X within male and female subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Mandy Chan, MBBS, Principal Investigator — The University of Hong Kong
Locations (1):
- Department of Medicine, Central, Hong Kong

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data